CLINICAL TRIAL: NCT04082832
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of Cu(II)ATSM in Patients With Amyotrophic Lateral Sclerosis/Motor Neuron Disease
Brief Title: CuATSM Compared With Placebo for Treatment of ALS/MND
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMD-2019-001
Record Dates: First submitted 2019-09-02; First posted 2019-09-09 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — copper (II) diacetyl-di(N(4)-methylthiosemicarbazone)

STUDY DESIGN:
Intervention Model Description: ANCOVA will be used to compare efficacy endpoints between CuATSM and placebo groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cu(II)ATSM (Active Comparator): Cu(II)ATSM Powder for Oral Suspension, 36 mg, to be reconstituted with Diluent (15 mL of sugar-free flavored pharmaceutical syrup) to provide an oral suspension for immediate consumption. Specified dose is 72 mg (2 bottles) taken fasting, before breakfast each day.
  Interventions: Drug: Cu(II)ATSM
- Placebo Powder for Oral Suspension (Placebo Comparator): Placebo Powder for Oral Suspension, to be reconstituted with Diluent (15 mL of sugar-free flavored pharmaceutical syrup) to provide an oral suspension for immediate consumption. Specified dose is 72 mg (2 bottles) taken fasting, before breakfast each day.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Cu(II)ATSM — oral suspension
  Arms: Cu(II)ATSM
Drug: Placebos — oral suspension
  Arms: Placebo Powder for Oral Suspension

SUMMARY:
Multicenter, randomized, double-blind, placebo controlled study to assess the tolerabilty and efficacy of CuATSM in patients with ALS/MND. Patients will be randomized 1:1 to CuATSM or placebo for 6 x 28-day cycles (24 weeks) of treatment.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to CuATSM or placebo for 6 x 28-day cycles (24 weeks) of treatment. Study drug is administered orally, once a day in fasted state (before breakfast). Assessments for safety (physical examination, vital signs, hematology, serum chemistry adverse events) will be conducted at baseline and following each cycle of treatment. Assessments for efficacy (Revised ALS Functional Rating Scale [ASLFRS-R] score, and Edinburgh Cognitive and Behavioral Amyotrophic Lateral Sclerosis Screen [ECAS] score, and seated slow vital capacity [SVC]) will be conducted at baseline and following 2, 4 and 6 cycles of treatment. Analysis of covariance (ANCOVA) will be used to compare efficacy endpoints between CuATSM and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* familial or sporadic ALS/MNS by Awaji-shima Consensus Recommendations
* not taking riluzole or on stable dose of riluzole for 4 weeks prior to screening visit
* no prior exposure to agents other than riluzole for treatment of ALS
* adequate bone marrow reserve, renal and liver function
* women of childbearing potential must have a negative pregnancy test and be non-lactating
* women and men with partners of childbearing potential must take effective contraception while on treatment

Exclusion Criteria:

* presence of a gastrointestinal disorder (eg, malabsorption) that might jeopardize intestinal absorption of study drug
* inability to perform seated SVC
* known immune compromising illness or treatment
* drug abuse or alcoholism
* clinically significant or active cardiovascular disease
* acute or chronic infection
* diagnosis of malignancy within 2 years prior to screening
* dementia that may affect patient understanding and/or compliance with study requirements and procedures
* current use of strong inducers or inhibitors of CYPs 2C19 and 2D6
* current us of medications (other than riluzole) that are metabolized predominantly by CYP 1A2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Revised ALS Functional Rating Scale (ALSFRS-R) total score (range: 48 [best] to 0 [worst]) | 24 weeks
  assessment of disease severity
Edinburgh Cognitive and Behavioral Amyotrophic Lateral Sclerosis Screen (ECAS) total score (range: 136 [best] to 0 [worst]) | 24 weeks
  assessment of cognitive function

SECONDARY OUTCOMES:
seated slow vital capacity (SVC) | 24 weeks
  assessment of respiratory function
rate of adverse events | 24 weeks
  tolerability assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Rowe, MD, Principal Investigator — Macquarie University
Locations (1):
- Macquarie University, Macquarie, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No